CLINICAL TRIAL: NCT02497690
Title: Effectiveness of Therapy Via Telemedicine Following Cochlear Implants
Acronym: TACIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); University of Colorado, Boulder (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 12-1103; 5U01DC013529 (NIH)
Record Dates: First submitted 2015-05-29; First posted 2015-07-14 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Congenital Sensorineural Deafness
Keywords: Cochlear Implant; Hearing Aid; Telemedicine
MeSH Terms: interventions — Telemedicine; Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- In-person ART (Active Comparator): In-person approach to provide ART.
  Interventions: Behavioral: In-person ART
- Telehealth ART (Experimental): Telemedicine technology approach (e.g. interactive video) to provide ART.
  Interventions: Behavioral: Telemedicine

INTERVENTIONS:
Behavioral: Telemedicine — Half of subjects will undergo six months of ART administered via telehealth. Therapy will be provided in the usual manner, except a computer will be used to facilitate the interaction.
  Other Names: Telehealth
  Arms: Telehealth ART
Behavioral: In-person ART — Half of subjects will undergo six months of ART administered in person. Therapy will be provided in the usual manner.
  Other Names: Standard of Care
  Arms: In-person ART

SUMMARY:
This study will assess the effectiveness of post-cochlear implant or hearing aid fitting Aural Rehabilitative Therapy (ART) delivered by means of telemedicine technology.

DETAILED DESCRIPTION:
Children with congenital sensorineural deafness can acquire relatively normal language if they undergo cochlear implantation surgery or hearing aid fitting followed by aural rehabilitation therapy in the first three to four years of life. High quality therapy, however, may not be available in many areas. This study will assess the effectiveness of post-cochlear implant or hearing aid fitting ART delivered by means of telemedicine technology. This will be accomplished primarily by evaluating subjects' language abilities using the 5th Edition of the Preschool Language Scales.

ELIGIBILITY:
Inclusion Criteria:

* been fitted with bilateral or unilateral cochlear implants, or bilateral hearing aids.
* focus on recruiting families who are members of minority groups.
* therapy must be provided in English.

Exclusion Criteria:

* the presence of one or more significant co-morbidities

  * blindness,
  * severe motor impairment,
  * autism,
  * significant genetic/chromosomal syndrome.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of subjects' language abilities. | 6 months
  Evaluation of subjects' language abilities will be conducted using the 5th Edition of the Preschool Language scales Preschool Language Scale (PLS-5)

CONTACTS AND LOCATIONS:
Overall Officials: James Grigsby, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States